CLINICAL TRIAL: NCT03240965
Title: Changes in Sensitivity of Swallowing-relevant Structures, Taste and Smell in Stroke Patients
Brief Title: Changes in Sensitivity, Taste and Smell in Stroke Patients
Acronym: 5S
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Tobias Braun, Principal Investigator, University of Giessen
Other Study IDs: GI-149/16
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dysphagia; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Volunteers <60 years: Volunteers, who are able to consent to participation in the study, as control.
  Interventions: Other: Sensitivity threshold; Diagnostic Test: Taste-/smell-test
- Volunteers >60 years: Volunteers, who are able to consent to participation in the study, as control.
  Interventions: Other: Sensitivity threshold; Diagnostic Test: Taste-/smell-test
- Stroke patients: Stroke patients with supratentorial stroke, who are able to consent to participation in the study.
  Interventions: Diagnostic Test: FEES (flexible endoscopic evaluation of swallowing); Other: Sensitivity threshold; Diagnostic Test: Taste-/smell-test; Diagnostic Test: Neuropsychological testing

INTERVENTIONS:
Diagnostic Test: FEES (flexible endoscopic evaluation of swallowing) — Endoscopical swallowing study in stroke patients only
  Groups: Stroke patients
Other: Sensitivity threshold — Determining sensitivity threshold using a pudendal electrode
Diagnostic Test: Taste-/smell-test — Taste-/smell-test
Diagnostic Test: Neuropsychological testing — Neuropsychological testing for neglect, agnosia
  Groups: Stroke patients

SUMMARY:
This study evaluates changes in swallowing using endoscopic swallowing studies and measuring of pharyngeal sensitivity, taste and smell in stroke patients. Younger (<60 years) and older (>60 years) volunteers will serve as control.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death. At least 50% of stroke patients develop dysphagia, leading to aspiration pneumonia, which is the main cause of death in stroke [2].

It is assumed that normal sensitivity is vital for aspiration-free swallowing and for the triggering of the swallowing reflex.

Ali et al. demonstrated aspiration-free swallowing in healthy volunteers who underwent local anaesthesia of oral and pharyngeal structures [1]. Power et al. showed a reduced sensitivity of pharyngeal structures in stroke patients prone to aspiration [3].

By combining measuring sensitivity and flexible endoscopic swallowing studies, this study further investigates the role of sensitivity in swallowing Neuropsychological deficits of swallowing, such as swallowing apraxia or buccal hemineglect, is assessed by neuropsychological testing.

Additionally, there is no systematic research investigating the change in smell and taste in correlation with changes in stroke patients

ELIGIBILITY:
Inclusion Criteria:

Volunteers:

* informed consent

Stroke patients:

* informed consent
* new supratentorial stroke (<72 hours old) confirmed by CT (computed tomography) or MRI (magnetic resonance imaging)

Exclusion Criteria:

* pre-existing stroke oder dysphagia
* extensive white matter lesions in CT- or MRI-scan
* allergies to odorous substances or flavoring
* contraindications for FEES (flexible endoscopic evaluation of swallowing), CT or MRI (stroke patients only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients are recruited in a university hospital's department of neurology.
  Volunteers >60years are recruited in a trauma surgery ward at the same university hospital.
  Volunteers <60 are recruited without specified characteristics (aside from in-/exclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dysphagia | 96 hours after initial symptoms
  Changes found in endoscopic swallowing study :
  Presence and severity of dysphagia (measured with Rosenbek's Penetration/Aspiration-scale)

SECONDARY OUTCOMES:
Neuropsychological deficits | 96 hours after initial symptoms
  Agnosia, neglect
Lesion site | 96 hours after initial symptoms
  Side, vascular territory, swallowing relevant structures
Sensitivity | 96 hours after initial symptoms
  Sensitivity of faucial pillar region
Taste/Smell | 96 hours after initial symptoms
  Smell-/Taste-score

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Braun, M.D., Principal Investigator — University Giessen
Locations (1):
- Universitätsklinikum Gießen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali GN, Laundl TM, Wallace KL, Shaw DW, Decarle DJ, Cook IJ. Influence of mucosal receptors on deglutitive regulation of pharyngeal and upper esophageal sphincter function. Am J Physiol. 1994 Oct;267(4 Pt 1):G644-9. doi: 10.1152/ajpgi.1994.267.4.G644. PMID 7943330
- [Background] Kidd D, Lawson J, Nesbitt R, MacMahon J. Aspiration in acute stroke: a clinical study with videofluoroscopy. Q J Med. 1993 Dec;86(12):825-9. PMID 8108539
- [Background] Power ML, Hamdy S, Singh S, Tyrrell PJ, Turnbull I, Thompson DG. Deglutitive laryngeal closure in stroke patients. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):141-6. doi: 10.1136/jnnp.2006.101857. Epub 2006 Sep 29. PMID 17012336
- [Derived] Braun T, Doerr JM, Peters L, Viard M, Reuter I, Prosiegel M, Weber S, Yeniguen M, Tschernatsch M, Gerriets T, Juenemann M, Huttner HB, Hamzic S. Age-related changes in oral sensitivity, taste and smell. Sci Rep. 2022 Jan 27;12(1):1533. doi: 10.1038/s41598-022-05201-2. PMID 35087097
- [Derived] Braun T, Hamzic S, Doerr JM, Peters L, Viard M, Reuter I, Prosiegel M, Weber S, Yenigun M, Tschernatsch M, Gerriets T, Juenemann M. Facilitation of oral sensitivity by electrical stimulation of the faucial pillars. Sci Rep. 2021 May 24;11(1):10762. doi: 10.1038/s41598-021-90262-y. PMID 34031508